CLINICAL TRIAL: NCT03707587
Title: A Phase II Study of M7824 in Subjects With Recurrent Respiratory Papillomatosis
Brief Title: M7824 in People With Recurrent Respiratory Papillomatosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Scott Norberg, D.O., Principal Investigator, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 190002; 19-C-0002
Record Dates: First submitted 2018-10-12; First posted 2018-10-16 (Actual); Results first posted 2020-10-14 (Actual); Last update posted 2022-09-29 (Actual); Status verified 2022-09

CONDITIONS: Recurrent Respiratory Papillomatosis; Respiratory Papillomatosis; Laryngeal Papilloma, Recurrent; Human Papilloma Virus
Keywords: Human Papilloma Virus (HPV); Monoclonal Antibody; PD-L1 Expression
MeSH Terms: conditions — Recurrent respiratory papillomatosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 1200 mg intravenous (IV) of M7824 (Experimental): Patients will receive 1200 mg intravenous (IV) of M7824 on day 1 of a 14 day cycle, every other week, for up to 12 weeks total treatment (6 cycles).
  Interventions: Drug: M7824

INTERVENTIONS:
Drug: M7824 — Patients will receive 1200 mg intravenous (IV) of M7824 on day 1 of a 14 day cycle, every other week, for up to 12 weeks total treatment (6 cycles).

SUMMARY:
Background:

Programmed cell death protein 1 (PD-L1) is a protein on the surface of cells. It regulates if a cell can be killed by immune system cells. It is thought to be able to affect the immune system response to diseased cells like those infected with a virus. The molecule M7824 interferes with the activity of PD-L1. It could help the immune system kill cells infected with a virus . Since recurrent respiratory papillomatosis is caused by a virus infection, this molecule could help.

Objective:

To see if M7824 works in treating recurrent respiratory papillomatosis.

Eligibility:

Adults ages 18 years or older with recurrent respiratory papillomatosis

Design:

Participants will be screened with:

Medical history

Physical exam

Blood and pregnancy tests

Endoscopy procedure in clinic. A small tube with a camera will look at the inside of the nose, throat, larynx, and upper windpipe.

Some participants will also be screened with a chest scan.

At the start of the study, participants will:

Have a sedated endoscopy procedure where biopsies will be taken.

Have blood tests.

Have apheresis. Blood will be collected by a tube in an arm vein. A machine will remove white blood cells. The rest of the blood will be returned into an arm vein.

Fill out a voice questionnaire.

Participants will get the study molecule into a vein over about 1 hour. They will get it every other week for up to 12 weeks.

Participants will repeat screening and starting procedures throughout the study. They will also review side effects and any medicine they are taking.

When they are done with the study treatment, participants will be evaluated by repeating the study procedures. They may be evaluated periodically until their disease progresses.

DETAILED DESCRIPTION:
Background

* Recurrent respiratory papillomatosis (RRP) is a rare papillomatous disease of the aerodigestive tract that is caused by the Human Papilloma Virus (HPV).
* RRP can progress to cause airway compromise, fatal pulmonary lesions, and invasive cancers.
* There is no effective systemic therapy for RRP. Patients typically require repeated interventional procedures for disease control.
* A recently completed phase II clinical trial investigating avelumab in subjects with aggressive RRP demonstrated an acceptable safety profile from Avelumab and a high rate of partial responses.
* RRP is characterized by frequent expression of PD-L1 and transforming growth factor beta (TGF)-beta in the tumor microenvironment.
* This clinical trial will evaluate the activity of M7824, a novel bifunctional fusion protein composed of a fully human Immunoglobulin G1 (IgG1) monoclonal antibody against human PD-L1 (avelumab) fused, via a flexible glycine-serine linker, to the soluble extracellular domain of human TGF- B receptor II (Transforming growth factor, beta receptor II (TGF-BRII), which functions as a TGF-B trap. This drug was selected for its demonstrated activity in a variety of cancers and for its acceptable safety profile.

Objective

- Determine the complete response rate for M7824 in the treatment of patients with RRP.

Eligibility

* Histologically confirmed diagnosis of RRP.
* One of the following:

  * A Derkay anatomic score of 10 or greater and a history of two or more endoscopic interventions in the last 12 months for control of RRP.
  * Pulmonary RRP with pulmonary disease that is measurable by computed tomography scan.
  * Tracheal involvement with RRP that has required either two or more endoscopic interventions in the last 12 months or a tracheostomy.
* Age 18 years or greater.
* Eastern Oncology Cooperative Group Performance Score of 0 or 1.

Design

* This is a phase II clinical trial with two cohorts that will enroll simultaneously.
* Cohort 1 will consist of subjects who have not been treated previously with an immune checkpoint inhibitor. Cohort 2 will consist of subjects whose disease has been treated previously with andrefractory to an immune checkpoint inhibitor. Each cohort will have a Simon optimal two-stage design with initial enrollment of 12 patients and expands 21 patients if one or more complete response(s) is/are observed in the initial patients. With amendment D, dated 7/24/2019, cohort 2 will be closed to further enrollment.

ELIGIBILITY:
* INCLUSION CRITERIA:

Recurrent Respiratory Papillomatosis (RRP) criteria:

* Histological diagnosis of RRP confirmed by pathology report from a Clinical Laboratory Improvement Amendments (CLIA)-certified laboratory.
* One of the following:

  * A Derkay anatomic score of 10 or greater and a history of two or more endoscopic interventions in the last 12 months for control of RRP.
  * Pulmonary RRP with pulmonary disease that is measurable by computed tomography scan and evaluated by Response Evaluation Criteria in Solid Tumors (RECIST) Criteria.
  * Tracheal involvement with RRP that has required either two or more endoscopic interventions in the last 12 months or a tracheostomy.
* Greater than or equal to 18 years of age.
* Able to understand and sign the Informed Consent Document.
* Clinical performance status of Eastern Cooperative Oncology Group (ECOG) 0 or 1.
* Willing to undergo endoscopic evaluation with biopsies in compliance with this protocol.
* No systemic therapy for RRP for at least 3 half-lives of the prior drug(s).
* Screening laboratory values must meet the following criteria and should be obtained within 14 days prior to first dose:

  * White Blood Count (WBC) > 2000/ microliter
  * Neutrophils > 1000/ microliter
  * Platelets > 75 x10(3)/ microliter
  * Hemoglobin > 9.0 g/dL
  * Serum Creatinine < 1.5 x upper limits of normal (ULN) OR estimated glomerular filtration rate (eGFR) > 30 mL/min (measured or calculated using the Modification of Diet in Renal Disease (MDRD) equation).
  * Aspartate aminotransferase (AST)/Alanine aminotransferase (ALT) less than or equal to 2.5 x ULN
  * Total Bilirubin: 1.5 x ULN
  * Prothrombin time (PT)/International Normalized Ratio (INR) and partial thromboplastin time (PTT) less than or equal to ULN
* Sexually active subjects (men and women) of reproductive potential must agree to use two methods of contraception: one highly effective and one other effective method throughout M7824 treatment and for at least 120 days after M7824 treatment. Highly Effective Methods are defined as: Intrauterine device (IUD), hormonal (birth control pills, injections, implants), tubal ligation and partner s vasectomy; Other are defined as: latex condom, diaphragm and cervical cap.
* Seronegative for human immunodeficiency virus (HIV) antibody. The experimental treatment being evaluated in this protocol depends on an intact immune system. Patients who are HIV seropositive can have decreased immune function and thus are likely less responsive to the experimental treatment.
* Seronegative for hepatitis B antigen, positive hepatitis B tests can be further evaluated by confirmatory tests (Hep B Deoxyribonucleic acid (DNA) Quant, hepatitis B virus (HBV) Viral Load), and if confirmatory tests are negative, the patient can be enrolled.
* Seronegative for hepatitis C antibody unless antigen negative. If hepatitis C antibody test is positive, then patients must be tested for the presence of antigen by Hep C Ribonucleic acid (RNA) Quant, hepatitis C virus (HCV) Viral Load and be HCV RNA negative.

EXCLUSION CRITERIA:

* Any severe acute or chronic medical or psychiatric conditions including recent (within the past year) or active suicidal ideation or behavior, liver disease, lung disease (with the exception of what is specified in inclusion criteria) , or laboratory abnormalities that, in the opinion of the investigators, may increase the risk associated with study participation or study drug administration, impair the ability of the subject to receive protocol therapy, or interfere with the interpretation of study results and in the judgment of the investigator, would make the patient inappropriate for entry into this study. Patients with mild to moderate asthma or chronic obstructive pulmonary disease (COPD) well controlled with oral or inhaled medications are permitted to enroll.
* Subjects with active, known or suspected autoimmune disease. Subjects with vitiligo, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, or psoriasis not requiring systemic treatment, are permitted to enroll.
* Subjects with a condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days of study drug administration. Inhaled, topical intranasal or intro-ocular steroids, and adrenal replacement doses <10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease.
* Prior organ transplantation, including allogeneic stem cell transplantation.
* Patients who are receiving any other investigational agents
* Pregnant or breast feeding. Women of childbearing potential must have a negative pregnancy test at screening. Women of childbearing potential include women who have experienced menarche and who have not undergone successful surgical sterilization (hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or are not postmenopausal. Post-menopause is defined as amenorrhea greater than or equal to 12 consecutive months. Note: women who have been amenorrheic for 12 or more months are still considered to be of childbearing potential if the amenorrhea is possibly due to prior chemotherapy, anti- estrogens, ovarian suppression or any other reversible reason.
* History of allergy to study drug components.
* History of severe hypersensitivity reaction to any monoclonal antibody (Grade greater than or equal to 3 National Cancer Institute (NCI)-Common Terminology Criteria for Adverse Events (CTCAE) v 5.0), any history of anaphylaxis, or uncontrolled asthma (that is, 3 or more features of partially controlled asthma).
* Clinically significant (i.e., active) cardiovascular disease: cerebral vascular accident/stroke (< 6 months prior to enrollment), myocardial infarction (< 6 months prior to enrollment), unstable angina, congestive heart failure (greater than or equal to New York Heart Association Classification Class II), or serious cardiac arrhythmia requiring medication.
* Persisting toxicity related to prior therapy of Grade >1 NCI-CTCAE v 5.0; however, alopecia, sensory neuropathy Grade less than or equal to 2 or other Grade less than or equal to 2 adverse events (AEs) not constituting a safety risk based on investigator's judgment are acceptable.
* Known alcohol or drug abuse.
* Vaccination within 4 weeks of the first dose of M7824 and 4 weeks after the last dose of M7824 are prohibited.
* Human papillomavirus (HPV) vaccination within one year of the first dose of M7824
* With amendment D, patients that received prior Programmed cell death protein 1 (PD-1) based immunotherapy will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2018-12-19 (Actual); Primary Completion 2019-10-29 (Actual); Study Completion 2022-07-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott Norberg, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Robbins Y, Friedman J, Clavijo PE, Sievers C, Bai K, Donahue RN, Schlom J, Sinkoe A, Hinrichs CS, Allen C, Abdul Sater H, Gulley JL, Norberg S. Dual PD-L1 and TGF-b blockade in patients with recurrent respiratory papillomatosis. J Immunother Cancer. 2021 Aug;9(8):e003113. doi: 10.1136/jitc-2021-003113. PMID 34462327
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2019-C-0002.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1 - Checkpoint Inhibitor Naive Patients: Patients with Recurrent Respiratory Papillomatosis (RRP) who are checkpoint inhibitor naïve will receive 1200 mg intravenous (IV) of M7824 on day 1 of a 14 day cycle, every other week.
- Cohort 2 - Patients Refractory to Checkpoint Inhibition: Patients with Recurrent Respiratory Papillomatosis (RRP) who are refractory to checkpoint inhibition will receive 1200 mg intravenous (IV) of M7824 on day 1 of a 14 day cycle, every other week.
Period: Overall Study
Arm/Group | Cohort 1 - Checkpoint Inhibitor Naive Patients | Cohort 2 - Patients Refractory to Checkpoint Inhibition
Started | 7 | 2
Completed | 7 | 1
Not Completed | 0 | 1
Not completed — Death | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 - Checkpoint Inhibitor Naive Patients | Cohort 2 - Patients Refractory to Checkpoint Inhibition | Total
Number analyzed (Participants) | 7 | 2 | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 1 | 8
  >=65 years | 0 | 1 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.42 (13.04) | 47.17 (16.32) | 39.79 (14.68)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 4
  Male | 4 | 1 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 7 | 1 | 8
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 5 | 1 | 6
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 7 | 2 | 9
Median Baseline Derkay Score [Median (Full Range); unit: scores on a scale] — The Derkay staging system incorporates an objective score based on the number of sites and bulkiness of papillomas within the pharynx, larynx and trachea, ranging from 0-3 for each site. The total score (combined value of the number of sites and bulkiness of papillomas within the pharynx, larynx and trachea) can range from 0 to 75. Higher values indicate worse disease.
  scores on a scale | 13 [2 to 24] | 13.5 [12 to 15] | 13 [2 to 24]

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Participants With a Complete Response
Description: Complete response for M7824 in the treatment of patients with RRP was assessed by the Response Evaluation Criteria in Solid Tumors (RECIST). Complete Response is defined as no evidence of papillomas on physical exam and/or clinic-based flexible nasopharyngolaryngoscopy and/or tracheoscopy or by exam under anesthesia (sedation or general anesthesia) with endoscopy and biopsies, and absence of disease by imaging if lesions are assessed by imaging.
Time Frame: Response was assessed by flexible endoscopy with or without imaging studies before treatment and 6 and 12 weeks after starting treatment.
Measure: Number; unit: proportion of participants
Arm/Group | Cohort 1 - Checkpoint Inhibitor Naive Patients | Cohort 2 - Patients Refractory to Checkpoint Inhibition
Number analyzed (Participants) | 7 | 2
proportion of participants | 0 | 0

2. Secondary Outcome: Number of Participants With a Partial Response
Description: Partial response for M7824 in the treatment of patients with RRP was assessed by the Response Evaluation Criteria in Solid Tumors (RECIST). Partial Response is defined as a decrease in Derkay anatomic score of 30 percent or greater, and a partial tumor response by imaging using RECIST 1.1 criteria.
Time Frame: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 - Checkpoint Inhibitor Naive Patients | Cohort 2 - Patients Refractory to Checkpoint Inhibition
Number analyzed (Participants) | 7 | 2
Participants | 1 | 0

3. Secondary Outcome: Number of Participants With ≥Grade 3 Adverse Events
Description: Adverse Events were assessed by the Common Terminology Criteria for Adverse Events (CTCAE v5.0). Grade 3 is defined as severe or medically significant but not immediately life-threatening. Grade 4 is defined as life-threatening consequences; urgent intervention indicated.
Time Frame: Per protocol, adverse events are documented from the first administration of the study therapy, Study Day 1, through 42 days after the study therapy was last administered, up to 24 weeks + 42 days.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 - Checkpoint Inhibitor Naive Patients | Cohort 2 - Patients Refractory to Checkpoint Inhibition
Number analyzed (Participants) | 7 | 2
Participants
  Grade 3 Dyspnea | 1 | 0
  Grade 3 Hypertension | 1 | 1
  Grade 3 Laryngeal obstruction | 4 | 1
  Grade 3 Lung infection | 1 | 0
  Grade 3 Pain | 1 | 0
  Grade 3 Sore throat | 1 | 1

4. Secondary Outcome: Number of Participants With Serious and Non-serious Adverse Events Assessed by the Common Terminology Criteria for Adverse Events (CTCAE v5.0)
Description: Here is the count of participants with serious and non-serious adverse events assessed by the Common Terminology Criteria for Adverse Events (CTCAE v5.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life-threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 - Checkpoint Inhibitor Naive Patients | Cohort 2 - Patients Refractory to Checkpoint Inhibition
Number analyzed (Participants) | 7 | 2
Participants | 7 | 2

ADVERSE EVENTS:
Time Frame: Per protocol, adverse events are documented from the first administration of the study therapy, Study Day 1, through 42 days after the study therapy was last administered, up to 24 weeks + 42 days. Beyond 42 days after the last administration (end of treatment), only adverse events which are serious and related to the M7824 need to be recorded until the patient is off study.
Arm/Group | Cohort 1 - Checkpoint Inhibitor Naive Patients | Cohort 2 - Patients Refractory to Checkpoint Inhibition
All-Cause Mortality (participants affected / at risk) | 0/7 | 1/2
Serious Adverse Events (participants affected / at risk) | 3/7 | 2/2
Other Adverse Events (participants affected / at risk) | 7/7 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 - Checkpoint Inhibitor Naive Patients (N=7) | Cohort 2 - Patients Refractory to Checkpoint Inhibition (N=2)
Laryngeal obstruction (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Lung infection (Infections and infestations) | 1 (1) | 0 (0)
Sudden death NOS (General disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 - Checkpoint Inhibitor Naive Patients (N=7) | Cohort 2 - Patients Refractory to Checkpoint Inhibition (N=2)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 2 (2)
Hypertension (Vascular disorders) | 4 (4) | 2 (3)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Laryngeal obstruction (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Lung infection (Infections and infestations) | 1 (1) | 0 (0)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) — ruptured umbilical cysts
Pain (General disorders) | 1 (1) | 0 (0)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 6 (12) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dry eye (Eye disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-12-01): https://cdn.clinicaltrials.gov/large-docs/87/NCT03707587/Prot_SAP_002.pdf
  • Informed Consent Form (2019-09-20): https://cdn.clinicaltrials.gov/large-docs/87/NCT03707587/ICF_001.pdf